CLINICAL TRIAL: NCT05010031
Title: Phase II Study to Examine Precision Radiation in Patients With Pathogenic Mutations in ATM
Brief Title: A Study of Reduced-dose Radiation in People With Metastatic Tumors With a Genetic Change
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-310
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Cancer
Keywords: Reduced-dose Radiation; Pathogenic Mutations; ATM (ataxia telangiectasia mutated); 21-310
MeSH Terms: conditions — Neoplasm Metastasis; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Intervention Model Description: Single arm, phase II noninferiority, prospective trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- radiation (Experimental): Subjects will receive reduced dose radiation to radiographically progressive lesions identified on imaging (including asymptomatic bone metastases).
  Interventions: Radiation: Palliative radiotherapy

INTERVENTIONS:
Radiation: Palliative radiotherapy — An initial cohort of 12 evaluable patients will be treated with 4Gyx2, with adaptive dosing planned for expansion cohorts pending the number of failures observed after 6 month observation of the initial cohort.

SUMMARY:
This study will test whether reduced-dose radiotherapy is an effective treatment for metastatic tumors with an ATM mutation. The researchers want to find the lowest dose of radiation that would still be effective to treat these tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy with at least one metastatic lesion referred for palliative radiotherapy
* Pathogenic mutation in ATM (somatic and germline allowed)
* ECOG performance status 0-2
* Age ≥ 18 years.
* Able to provide informed consent.
* Patients at reproductive potential must agree to practice an effective contraceptive method during radiation treatments.
* Expected life expectancy of at least 6 months

Exclusion Criteria:

* Previous radiotherapy to the intended treatment site that precludes developing a treatment plan that respects normal tissue tolerances.
* Serious medical co-morbidities precluding radiotherapy.
* Pregnant or breast-feeding women.
* Lesions excluded from de-escalation include regions in which the risk of local disease progression is unacceptably high, including CNS disease and cord compression, and areas in which re-irradiation would not be feasible, including spinal cord overlap.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Treatment failure rate of irradiated lesion | 6 month
  Defined as (i) radiographic progression or (ii) re-irradiation to the treated site. If PET is performed, radiographic criteria will be evaluated per PERCIST

CONTACTS AND LOCATIONS:
Overall Officials: Amy Xu, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/